CLINICAL TRIAL: NCT07063836
Title: Management of Compromised Adjacent Extraction Sockets Via Vestibular Socket Therapy Versus Early Contour Augmentation a Randomized Controlled Clinical Trial
Brief Title: Management of Multiple Adjacent Extraction Sockets
Acronym: VST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25-026
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Dental Implant in Compromised Adjacent Sockets
Keywords: dental implant, compromised socket, bone augmentation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vestibular socket therapy (Experimental): A small incision (1 cm) is made on (vestibular area) near the base of the extracted teeth, extending slightly towards neighboring teeth. This creates a pouch for accessing the socket and surrounding bone.An immediate implant is inserted using a guide and covered with a cortical membrane
  Interventions: Procedure: VST
- Contour augmentation and early implant placement (Active Comparator): early implant placement after socket healing for four weeks using bioplug along with contour augmentation using bone and membrane
  Interventions: Procedure: contour augmentation and early implant placement

INTERVENTIONS:
Procedure: VST — atraumatic extraction to the hopeless teeth will be performed using periotomes followed by conventional forceps under local anesthesia.A small incision (1 cm) is made on (vestibular area) near the base of the extracted teeth, extending slightly towards neighboring teeth.Using special instruments from the VST kit, the gum tissue is carefully dissected to expose the underlying bone and an immediate implant is placed using a surgical guide. the augmentation is done using A mixture of bone chips harvested from the surgical site (autogenous bone) and a bone-grafting material (deproteinized bovine bone mineral) is used to fill any gaps and support the implant, especially in the labial bone wall (labial plate).
  A special 0.6 mm thick membrane is inserted through the access incision. the vestibular incision is then sutured and the provisional is inserted.
  Arms: vestibular socket therapy
Procedure: contour augmentation and early implant placement — Teeth extraction : minimally invasive adjacent teeth extraction under anesthesia using periotome and forceps.
  the empty sockets will be filled with a special collagen material (BioPlug) to aid healing for 4 to 8 weeks.
  flap elevation : a full-thickness flap will be carefully raised using a crestal incision extended one tooth mesial and distal to the extraction location, then connected with two vertical incisions extended through the sulcus forming a trapezoid flap.
  Implants Insertion: The two implant is then placed into the prepared sockets using surgical guide.
  Bone Grafting: Any bone deficiencies are addressed by grafting. This involves placing a layer of (autogenous bone) directly on the two implants' surface, followed by a layer of a bone-grafting material (Demineralized Bone Matrix).
  Membrane Placement: A double-layered collagen membrane is used to cover the grafted area.
  Flap Closure: The previously lifted flap is repositioned and sutured back in place.
  Arms: Contour augmentation and early implant placement

SUMMARY:
While early implant placement with guided bone regeneration (GBR) offers advantages, the desire for reduced treatment time and fewer surgical steps continues to drive the exploration of alternative approaches. In this context, the recent introduction of vestibular socket therapy (VST) presents an intriguing option. VST utilizes a minimally invasive tunnel access technique through the vestibular area to perform socket augmentation for immediate implant placement in compromised extraction sockets .

DETAILED DESCRIPTION:
The concept of immediate implant placement has been around for a while. Professor Wilfried Schulte conducted the first study on this technique in 1978, Extensive studies conducted over the past 40 years have demonstrated that immediate implant placement is a safe and effective method for restoring teeth that are badly destructed.

While immediate implant placement has been shown as a viable option, new studies using advanced imaging techniques (cone beam CT scans) reveal limitations in the front upper jaw (anterior maxilla).

Thin Bone Walls: These scans show that a thick bone wall, ideal for implant stability, is uncommon in this area. Only about 5% of patients have a thick wall (>1mm) in the central incisor region.

Facial Bone Defects: Another recent study found that over half (52%) of implant sites in the central incisor area have a missing facial bone wall (defect).

These findings highlight the main concerns with immediate implants in the front upper jaw:

Bone Instability: Thin bone and missing facial bone can lead to an unstable implant, especially in the thin tissue layer at the front of the jaw (labial plate).

Soft Tissue instability: An unstable implant can cause the gum tissue to recede, compromising the cosmetic outcome in this highly visible area.

researchers like Buser et al. propose a treatment option that offers documented long-term predictability for achieving good aesthetic outcomes. This approach involves:

Early Implant Placement (Type 2): The implant is placed shortly after tooth extraction.

Flap Surgery: This surgical technique allows for better access to the bone for grafting.

Guided Bone Regeneration: Bone grafting material is used to stimulate new bone growth in the missing facial bone area.

Submerged Healing: The implant is left covered by gum tissue for a period of healing before attaching the final restoration.

This alternative approach addresses the challenges of immediate implant placement in cases with missing facial bone walls in the front upper jaw, while offering a predictable and aesthetically pleasing long-term solution.

A recent studies compared an alternative approach to the contour augmentation technique. The technique is the novel vestibular socket therapy proposed by ELaskary et al.

The findings suggest VST may be a viable option for these situations, offering comparable bone formation and improved soft tissue stability while streamlining the treatment process with fewer surgical interventions.

The study found that VST offered several advantages:

More stable gum tissue Similar bone growth compared to contour augmentation Faster treatment time Fewer surgeries Overall, VST appears to be a promising alternative to contour augmentation for implant placement.

ELIGIBILITY:
Inclusion Criteria:

- patients with two adjacent hopeless maxillary teeth or remaining roots in the esthetic region missing coronal tooth structure, type II socket (deficient labial plate of bone and intact overlying soft tissues), adequate palatal bone, ≥ 3 mm apical bone to engage the immediately placed implants, thereby achieving optimum primary stability (a minimum of 30 Ncm insertion torque) following teeth extraction.

acceptable compliance and oral hygiene.

Exclusion Criteria:

medically compromised patients. (Systemic diseases). general contraindication for implant placement. (Untreated periodontitis, severe bruxism , immunosuppression , uncontrolled diabetes , smokers , patients under radiation therapy, patients on bisphosphonate medications).

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
soft tissue stability | 6 months after final restoration
  it will be measured digitally using the intraoral scanner. A preoperative scanning, immediate postoperative, 3 months postoperative and 6 months postoperative scanning will be done.

SECONDARY OUTCOMES:
buccal plate of bone regeneration | 6 months
  measuring the thickness of the labial plate of bone. It will be measured preoperatively, immediate postoperative to measure the amount of the augmented bone, 3 months postoperatively and 6 months post operative. Tool to be used: cone beam computed tomography (cbct)

OTHER OUTCOMES:
Pink esthetic score | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Yousef, B.D.S, Principal Investigator — British University In Egypt
Locations (1):
- The British university in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No